CLINICAL TRIAL: NCT01697696
Title: A Multi-center, Randomized, Double-blind, 52-week Study to Assess the Safety of NVA237 Compared to QAB149 in Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Have Moderate to Severe Airflow Limitation
Brief Title: Long Term Safety Study of NVA237 vs QAB149 in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2319; 2012-002728-34 (EudraCT Number)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, NVA237, QAB149, glycopyrronium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 dose 1 (Experimental): NVA237 dose 1
  Interventions: Drug: NVA237
- Long-acting beta 2-agonist (LABA) (Active Comparator): QAB149
  Interventions: Drug: Long-acting beta 2-agonist (LABA); Drug: Placebo

INTERVENTIONS:
Drug: NVA237 — NVA237 will be supplied in capsule form in blister packs for use in the Novartis Concept 1 SDDPI
  Arms: NVA237 dose 1
Drug: Long-acting beta 2-agonist (LABA) — QAB149 and matching placebo will be supplied in capsule form in blister packs for use in the Novartis Concept 1 SDDPI
  Arms: Long-acting beta 2-agonist (LABA)
Drug: Placebo — Placebo to match QAB149
  Arms: Long-acting beta 2-agonist (LABA)

SUMMARY:
The purpose of the study is to provide long term safety data of NVA237. This study will assess the safety and tolerability of a single dose strength of NVA237.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with COPD according to GOLD 2011 who have signed informed consent.
2. Patients with airflow limitation of 30-80% post-bronchodilator FEV1 at run-in.
3. Current or ex-smokers with a smoking history of at least 10 pack years
4. Patients with a mMRC score of at least 2 at run-in.

Exclusion Criteria:

1. Patients contraindicated for muscarinic antagonist agents and beta-2 agonists
2. Patients with a history of malignancy of any organ system, treated or untreated, within the last five years
3. Patients with narrow-angle glaucoma, BPH or bladder-neck obstruction or moderate-severe renal impairment or urinary retention
4. Patients who had a COPD exacerbation within 6 weeks prior to screening.
5. Patients requiring long term oxygen therapy prescribed for more than 12 hr per day.
6. Patients with a history of asthma.
7. Patients with an onset of respiratory symptoms, including COPD diagnosis, prior to 40 years of age.
8. Patients with a blood eosinophil count of greater than 600 mm/3 during run-in
9. Patients with concomitant pulmonary disease
10. Patients with a history of certain cardiovascular co-morbid conditions
11. Patients with a diagnosis of alpha-1 anti-trypsin deficiency
12. Patients with active pulmonary tuberculosis
13. Patients in the active phase of a pulmonary rehabilitation programme
14. Other protocol-defined inclusion / exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (55):
  - Novartis Investigative Site, Gulf Shores, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Glastonbury, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Oakland Park, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Couer D'Alene, Idaho
  - Novartis Investigative Site, Newburgh, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Florence, Kentucky
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Biddeford, Maine
  - Novartis Investigative Site, Worchester, Massachusetts
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Fremont, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Calabash, North Carolina
  - Novartis Investigative Site, Tabor City, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Zanesville, Ohio
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Warwick, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, North Myrtle Beach, South Carolina
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Kingwood, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, White River Junction, Vermont
  - Novartis Investigative Site, Burke, Virginia
  - Novartis Investigative Site, Fredericksburg, Virginia
  - Novartis Investigative Site, Manassas, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Oregon, Wisconsin

REFERENCES:
- [Derived] Mahler DA, Gifford AH, Satti A, Jessop N, Eckert JH, D'Andrea P, Mota F, Banerjee R. Long-term safety of glycopyrrolate: A randomized study in patients with moderate-to-severe COPD (GEM3). Respir Med. 2016 Jun;115:39-45. doi: 10.1016/j.rmed.2016.03.015. Epub 2016 Mar 22. PMID 27215502

RESULTS

PARTICIPANT FLOW:
Groups:
- NVA237: 12.5 μg twice-daily
- QAB149: 75 μg once-daily
Period: Overall Study
Arm/Group | NVA237 | QAB149
Started | 254 | 257
Safety Set | 251 | 256 (Safety set included a patient that was treated, but not randomized)
Full Analysis Set (FAS) | 251 | 255
Completed | 207 | 210
Not Completed | 47 | 47
Not completed — Study terminated by sponsor | 0 | 3
Not completed — Protocol deviation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 10 | 7
Not completed — Subject/guardian decision | 31 | 35

BASELINE CHARACTERISTICS:
Population: The Safety set included all patients that received at least one dose of study drug and had at least one-post baseline assessment . Subjects were analyzed according to the treatment they received (if a subject incorrectly took more than one treatment, the subject was analyzed according to the treatment they were randomized to).
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 | QAB149 | Total
Number analyzed (Participants) | 251 | 256 | 507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.15) | 63.2 (8.91) | 63.3 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 107 | 217
  Male | 141 | 149 | 290

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Safety and Tolerability in Terms of Adverse Event (AE) Reporting Rate
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal lab finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgments of the investigators represent significant hazards.
Time Frame: 52 weeks
Population: Safety population - all patients who received at least one dose of study drug whether or not they were randomized. Only patients with safety assessments were included in this analysis
Measure: Number; unit: Percentage of participants
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 251 | 256
Percentage of participants | 77.3 | 77

2. Secondary Outcome: Time to Treatment Discontinuation
Description: Discontinuation rates are calculated using the Kaplan Meier method. The protocol allowed patients to discontinue outside the treatment window, hence we have a patient who discontinued at Day 388. Reasons for discontinuing treatment are Subject/guardian decision, Adverse event, Protocol deviation Lack of efficacy, Physician decision, Dosing error, Disease improvement under study, Pregnancy, Technical problems
Time Frame: 52 Weeks
Population: The Safety set consisted of all patients that received at least one dose of study medication and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 251 | 256
Days | NA [NA to NA] — NA - Insufficient number of participants with events | 388 [388 to NA] — NA - Insufficient number of participants with events

3. Secondary Outcome: Change From Baseline in Mean Forced Expiratory Volume (Average of the Two FEV1 Measurements 45 and 15 Minutes Pre-dose) in One Second at Week 52
Description: Change from baseline in pre-dose trough FEV1 was analyzed using a repeated measures analysis of covariance model which contained treatment, baseline FEV1, visit, baseline smoking status, baseline ICS use, COPD severity and treatment by visit, visit by baseline FEV1 interactions. An unstructured variance-covariance error matrix was used .Pulmonary function assessments were performed using centralized spirometry according to international standards. Pre-dose trough FEV1 was defined as the mean of FEV1 at -45 min and -15 min before the morning dose at Week 52. Baseline FEV1 was defined as the mean of the pre-dose FEV1 at -45 min and -15 min on Day 1.
Time Frame: -45 min and -15 minutes baseline and at Week 52
Population: The Full Analysis set (FAS) included patients who received at least one dose of study medication. Patients were analyzed according to the treatment to which they were randomized. Only participants from the full analysis set, who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 229 | 227
Liters | 0.056 (0.0211) | 0.060 (0.0213)

4. Secondary Outcome: Change From Baseline in Pre-dose Forced Expiratory Volume (FEV1) in One Second at All Post Baseline Timepoints
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1.
Time Frame: -45 min and -15 minutes baseline and at Week 52
Population: The Full Analysis set (FAS). At each day/time point, only subjects with a value at both baseline and the respective day/time point are included. Only participants with baseline and specific post baseline time points were included in the analysis for that time point.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 229 | 227
Liters
  Day 29/-45min | 0.104 (0.1848) | 0.118 (0.2093)
  Day 29/-15min | 0.123 (0.1872) | 0.138 (0.2061)
  Day 57/-45min | 0.098 (0.2017) | 0.101 (0.2091)
  Day 57/-15min | 0.120 (0.2025) | 0.107 (0.2111)
  Day 85/-45min | 0.105 (0.2410) | 0.085 (0.2255)
  Day 85/-15min | 0.111 (0.2137) | 0.099 (0.2328)
  Day 141/-45min | 0.071 (0.2168) | 0.089 (0.2595)
  Day 141/-15min | 0.096 (0.2060) | 0.108 (0.2670)
  Day 197/-45min | 0.071 (0.2370) | 0.082 (0.2637)
  Day 197/-15min | 0.073 (0.2150) | 0.090 (0.2827)
  Day 253/-45min | 0.092 (0.2774) | 0.087 (0.2679)
  Day 253/-15min | 0.094 (0.2100) | 0.103 (0.2659)
  Day 309/-45min | 0.068 (0.2850) | 0.094 (0.2594)
  Day 309/-15min | 0.088 (0.2845) | 0.112 (0.2638)
  Day 365/-45min | 0.057 (0.2541) | 0.088 (0.2521)
  Day 365/-15min | 0.087 (0.2592) | 0.090 (0.2627)

5. Secondary Outcome: Change From Baseline in Pre-dose Forced Vital Capacity (FVC) at All Post-baseline Timepoints
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FVC was defined as the average of the pre-dose FVC measured at -45 minutes (min) and -15 min at day 1.
Time Frame: -45 min and -15 minutes baseline and at Week 52
Population: Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Only participants with baseline and specific post baseline time points were included in the analysis for that time point.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 229 | 227
Liters
  Day 29/-45min | 0.191 (0.3433) | 0.170 (0.3536)
  Day 29/-15min | 0.217 (0.3440) | 0.194 (0.3495)
  Day 57/-45min | 0.168 (0.3501) | 0.140 (0.3655)
  Day 57/-15min | 0.210 (0.3414) | 0.178 (0.3610)
  Day 85/-45min | 0.171 (0.3907) | 0.094 (0.3711)
  Day 85/-15min | 0.188 (0.3875) | 0.118 (0.3823)
  Day 141/-45min | 0.159 (0.3742) | 0.112 (0.3822)
  Day 141/-15min | 0.182 (0.3706) | 0.141 (0.4068)
  Day 197/-45min | 0.140 (0.3879) | 0.075 (0.4043)
  Day 197/-15min | 0.133 (0.3992) | 0.083 (0.4183)
  Day 253/-45min | 0.167 (0.4567) | 0.100 (0.4219)
  Day 253/-15min | 0.153 (0.3703) | 0.125 (0.3984)
  Day 309/-45min | 0.120 (0.4539) | 0.094 (0.4122)
  Day 309/-15min | 0.149 (0.4451) | 0.114 (0.4207)
  Day 365/-45min | 0.116 (0.4053) | 0.109 (0.4426)
  Day 365/-15min | 0.143 (0.3970) | 0.097 (0.4171)

6. Secondary Outcome: Change From Baseline in COPD Symptoms
Description: The total symptom score was defined as the sum of individual cores for respiratory symptoms, cough, wheeze, amount of sputum, color of sputum, and reathlessness. Where a patient had a morning score and an evening score for an individual symptom on one particular day then the worst score was to be taken as the daily score for that symptom. Each symptom scale ranged from 0-3 where 0 was no symptoms and 3 was the worst. The total daily/daytime/nighttime symptom score consists of looking at the score for 6 symptoms and can therefore have a minimum score of 0 or a maximum of 18.
Time Frame: 52 weeks
Population: Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Only participants from the full analysis set, who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed."
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 251 | 255
scores on a scale
  Daily total symptom score (n=231, 227) | -1.18 (0.137) | -1.47 (0.137)
  Daytime total symptom score (n=221, 220) | -0.95 (0.129) | -1.14 (0.129)
  Nighttime total symptom score (n=226, 222) | -1.11 (0.126) | -1.25 (0.128)

7. Secondary Outcome: Change From Baseline in COPD Symptoms
Description: Percentage of days with 'no daytime symptoms' A day with 'no daytime symptoms' was defined from the diary data as any day where the patient had recorded in the evening no cough, no wheeze, no production of sputum and no feeling of breathlessness (other than when running) and no puffs of rescue medication during the past 12 hours (approximately 8 am to 8pm). However, a patient was not considered symptom free if they had used rescue medication that day even if his/her total daytime symptoms score was zero. Percentage of nights with 'no nighttime awakenings' A night with 'no nighttime awakenings' was defined from diary data as any night where the patient did not wake up due to symptoms. The total number of nights with 'no nighttime awakenings' over the treatment period was divided by the total number of nights where diary recordings had been made in order to derive the percentage nights with 'no nighttime awakenings'.
Time Frame: 52 weeks
Population: Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Only participants from the full analysis set, who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days / nights
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 251 | 255
Percentage of days / nights
  Nights with no nighttime awakenings (n=226, 222) | 17.4 (1.84) | 18.0 (1.86)
  Days with no daytime symptoms (n=221, 220) | 6.0 (1.38) | 5.1 (1.38)
  Days able to perform daily activities(n=221,220) | 5.4 (2.09) | 8.5 (2.10)

8. Secondary Outcome: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication
Description: The number of puffs of rescue medication taken in the previous 12 hours was recorded by the patients in the eDiary in the morning and evening. The total number of puffs of rescue medication per day over the 52 week treatment period was calculated and divided by the total number of days with non-missing rescue data to derive the mean daily number of puffs of rescue medication taken for the patient. If the number of puffs was missing for part of the day (either morning or evening), then a half day was used in the denominator. Change from baseline in number of puffs were analyzed using a linear mixed model which contained treatment, baseline number of puffs, baseline smoking status, baseline ICS use and COPD disease severity as fixed effects with center as a random effect
Time Frame: 52 weeks
Population: Only participants from the full analysis set, who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 251 | 255
Number of puffs
  Daily (n=231, 227) | -1.16 (0.199) | -1.79 (0.199)
  Daytime (n=221, 220) | -0.71 (0.112) | -1.05 (0.112)
  Nighttime (n=226, 222) | -0.52 (0.094) | -0.73 (0.095)

9. Secondary Outcome: Time to First COPD Exacerbation (Moderate or Severe).
Description: COPD exacerbations are considered to be moderate if treatment with systemic corticosteroids and/or antibiotics was required. COPD exacerbations are considered to be severe if hospitalizations were required. Rates are calculated using the Kaplan Meier method.
Time Frame: 52 weeks
Population: The Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Patients were analyzed according to the treatment to which they were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NVA237 | QAB149
Number analyzed (Participants) | 251 | 255
Days | NA [NA to NA] — NA - Insufficient number of participants with events | NA [NA to NA] — NA - Insufficient number of participants with events

ADVERSE EVENTS:
Arm/Group | NVA237 | QAB149
Serious Adverse Events (participants affected / at risk) | 33/251 | 34/256
Other Adverse Events (participants affected / at risk) | 165/251 | 170/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=251) | QAB149 (N=256)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2
ANGINA PECTORIS (Cardiac disorders) | 1 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 1
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 2 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 5 | 4
SEPSIS (Infections and infestations) | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 1
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
CEREBRAL THROMBOSIS (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 1
DYSARTHRIA (Nervous system disorders) | 0 | 1
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 1 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1
ALCOHOLISM (Psychiatric disorders) | 0 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 1
DYSPHORIA (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 11 | 12
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1
AORTIC DISSECTION (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=251) | QAB149 (N=256)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 3
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 2
DENTAL CARIES (Gastrointestinal disorders) | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 9 | 5
DRY MOUTH (Gastrointestinal disorders) | 3 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 3
NAUSEA (Gastrointestinal disorders) | 9 | 6
TOOTHACHE (Gastrointestinal disorders) | 3 | 4
VOMITING (Gastrointestinal disorders) | 5 | 7
FATIGUE (General disorders) | 11 | 3
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 3
OEDEMA PERIPHERAL (General disorders) | 2 | 6
SEASONAL ALLERGY (Immune system disorders) | 1 | 3
BRONCHITIS (Infections and infestations) | 11 | 9
DIVERTICULITIS (Infections and infestations) | 2 | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 3 | 2
INFLUENZA (Infections and infestations) | 7 | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 10
NASOPHARYNGITIS (Infections and infestations) | 20 | 27
ORAL CANDIDIASIS (Infections and infestations) | 1 | 5
RHINITIS (Infections and infestations) | 5 | 1
SINUSITIS (Infections and infestations) | 10 | 12
TOOTH ABSCESS (Infections and infestations) | 3 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 | 16
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 10 | 5
URINARY TRACT INFECTION (Infections and infestations) | 8 | 5
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 | 12
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 4 | 2
CONTUSION (Injury, poisoning and procedural complications) | 4 | 0
FALL (Injury, poisoning and procedural complications) | 5 | 3
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 3 | 4
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 4
BLOOD PRESSURE INCREASED (Investigations) | 4 | 1
WEIGHT DECREASED (Investigations) | 3 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 2
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 6
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 3
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 3 | 0
DIZZINESS (Nervous system disorders) | 5 | 6
HEADACHE (Nervous system disorders) | 4 | 8
SYNCOPE (Nervous system disorders) | 4 | 1
TREMOR (Nervous system disorders) | 4 | 2
ANXIETY (Psychiatric disorders) | 4 | 7
DEPRESSION (Psychiatric disorders) | 3 | 4
INSOMNIA (Psychiatric disorders) | 4 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 4
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 83 | 88
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 | 20
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 | 9
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 9 | 9
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 11 | 11
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 3
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 5
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 | 6
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 3 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 5 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 3
HYPERTENSION (Vascular disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety